CLINICAL TRIAL: NCT06792396
Title: Study to Understand the Diagnostic Measures, Management Options and Long Term Outcomes in a Local Cohort of Patients with Electrical Status Epilepticus in Sleep, Also Known As a Developmental And/or Epileptic Encephalopathy with Spike-Wave Activation in Sleep
Brief Title: Study of Patients with Electrical Status Epilepticus in Sleep
Acronym: SPESES
Status: Recruiting | Type: Observational
Sponsor: East Suffolk and North Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 23/213
Record Dates: First submitted 2024-12-30; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Electrical Status Epilepticus in Sleep

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Our aims are:

1. To understand the diagnostic practices, treatment and long term management and outcomes for patients diagnosed with ESES locally.
2. To establish a regional and national guideline for the diagnosis and management of patients with ESES.

The secondary questions that can be addressed with this case series review include the variability of clinical care given to patients with this condition, and for example, the duration of time it takes to obtain diagnostic tests and assessments by psychologists.

DETAILED DESCRIPTION:
The Paediatric consultants specialising in epilepsy and neurodisability at ESNEFT that are on the delegation log will identify patients who have been diagnosed with ESES since 2010.

This list of patients will be pseudo-anonymised (by tagging patients with a random identification number). Patient identifiable data including local hospital identification number and date of birth will be collected on the local case record form (CRF) to enable retrospective data collection. The hospital number will remain within the Trust, meaning only the local NHS staff responsible for care have access to personal identifying information.

No personal data will be leaving ESNEFT. Patients will be identified by their treating clinicians who are aware of their diagnoses and will list the patient hospital number in a password-protected spreadsheet. The list will be pseudo-anonymised by assigning a random number to the case, and anonymised data will be then gathered in the data collection tool. This ensures patient confidentiality. We will use two separate spreadsheets, one documenting the patient's hospital number and their assigned study number. This spreadsheet will not contain any other identifiable patient details (i.e. patient name, age, date of birth etc). A separate spreadsheet will contain patient study numbers only with medical history information relevant to the study. Both will be password protected secured on the NHS site. All data will be entered promptly and frequently cleaned.

The patient electronic patient records will be mined for information regarding age at onset, symptoms at onset, developmental issues, ongoing clinical history- recorded as Human Phenotype Ontology terms, diagnostic tests, duration of time till diagnostic tests such as electroencephalography in sleep or genetic tests undertaken, and duration of time till neuropsychology assessments (if any) undertaken. We will also record the underlying cause for ESES (where available), whether the patient has been discharged from ongoing follow-up and if there are ongoing physical or neuropsychological issues, at their current age. This information will be collected using a data collection tool, which will be an excel spreadsheet.

The anonymised dataset will be analysed by the research team. We will involve patient and family groups in the review of documents prior to dissemination of research findings.

ELIGIBILITY:
Inclusion Criteria:

1. Any Paediatric patient (up to 16 years old) who has been managed for electrical status epilepticus in sleep or developmental and/or epileptic encephalopathy with spike-wave activation in sleep, by clinicians at East Suffolk and North Essex NHS Foundation Trust, within the last 15 years.
2. Patients meeting criteria 1) with available electronic health records.

Exclusion Criteria:

1. Any Paediatric patient (up to 16 years old) with epilepsy managed by clinicians at East Suffolk and North Essex NHS Foundation Trust, where the diagnosis of electrical status epilepticus in sleep or developmental and/or epileptic encephalopathy with spike-wave activation in sleep was not confirmed.
2. Patients without electronic health record availability.
3. Patients over 16 years old.
4. Patients who have opted out of data use as per national opt out policy.

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Within the East Suffolk and North Essex region
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Creation of an evidence-based guideline | Over the past 10-15 years
  The primary outcome measure for the study is the creation of an evidence-based guideline using clinical experience of managing patients with electrical status epilepticus in sleep.

SECONDARY OUTCOMES:
Diagnosis criteria | Over the last 10-15 years
  Diagnostic criteria used when patients were given a diagnosis of electrical status epilepticus in sleep (ESES)
Treatments used | Over the last 10-15 years
  Treatments used prior to and after diagnosis of ESES
Treatment response monitoring | Over the last 10-15 years
  How treatment response was monitored
Duration of time | Over the last 10-15 years
  Duration of time taken to assess a patient using electroencephalography and neuropsychological tests
Long term outcomes and clinical spectrum | Over the last 10-15 years
  Long term outcomes and clinical spectrum associated with ESES

CONTACTS AND LOCATIONS:
Locations (1):
- East Suffolk and North Essex NHS Foundation Trust, Colchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No